CLINICAL TRIAL: NCT05296954
Title: Localization of Anatomical Structures Involved in Nodal Tachycardias by High Density Mapping. Feasibility Study.
Brief Title: Localization of Anatomical Structures Involved in Nodal Tachycardias by High Density Mapping.
Acronym: KOCH-MAPPING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/21/0076
Record Dates: First submitted 2022-03-04; First posted 2022-03-25 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Atrioventricular Nodal Reentry Tachycardia; Supraventricular Tachycardia
Keywords: Voltage mapping; Atrioventricular node mapping
MeSH Terms: conditions — Tachycardia, Atrioventricular Nodal Reentry; Tachycardia, Supraventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Tachycardia
  Interventions: Procedure: high resolution cartography
- Group 2 (Active Comparator): Without tachycardia
  Interventions: Procedure: high resolution cartography

INTERVENTIONS:
Procedure: high resolution cartography — High-resolution electro-anatomical mapping will be performed in each group with the RHYTHMIA HDx system to obtain an activation and voltage map of the Koch triangle and surrounding areas.

SUMMARY:
The aim of the present work is to analyze the capacity of high resolution mapping systems to determine the precise location of the AV node and peri-nodal slow-conducting pathways, using standard recording parameters, but also off-line additional filter changes and additional techniques (conduction velocities, isochrones and dV/dt). The investigative team plan a prospective monocentric study.

Detailed high resolution mapping of the Koch triangle and neighboring areas will be collected through the RHYTHMIA HDx 3D electro-anatomical mapping system and the multipolar ORION catheter. This sample will consist of 2 groups of patients: the first will include patients referred for AVNRT ablation and the second will include control patients (without AVNRT), referred for another indication requiring similar mapping system. If visualized, position of the slow pathway and AV node will be compared with the ablation areas, which will be set conventionally under fluoroscopy.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Patients without heart disease presenting with reciprocal tachycardia by intra-nodal reentry.

Group 2: Control subjects, without nodal tachycardia, without heart disease, and admitted for ablation of atrial fibrillation or ventricular extrasystoles on a healthy heart and with a 3D system.

Exclusion Criteria:

* Presence of underlying structural heart disease or history of atrial ablation or atrial tachycardia
* Minor or protected patient
* Patient under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Determine the precise location of the AV node | 7 months
  Determine the precise location of the AV node with off-line additional filter changes and additional techniques (conduction velocities, isochrones and dV/dt).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MAURY, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No